CLINICAL TRIAL: NCT02513030
Title: Cardioverter Defibrillator Replacement With Induction of Ventricular Fibrillation and Defibrillation Testing
Acronym: SIMPLER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Michael Glikson, Director of Davidai Arrhythmia Center, Sheba Medical Center
Other Study IDs: SHEBA-15-2033-MG-CTIL
Record Dates: First submitted 2015-03-05; First posted 2015-07-31 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Defibrillation Capacity of Defibrilators After Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Replacement of defibrillator
  Interventions: Procedure: Defibrillation testing during ICD replacement

INTERVENTIONS:
Procedure: Defibrillation testing during ICD replacement

SUMMARY:
The SIMPLE study was a large one, and lasted quite a few years due to its design as a randomized controlled trial and the follow up needed to reach an endpoint. The investigators aim to conduct an observational pilot study looking at frequency of positive findings during VF testing . The comparator will be the rate of findings during testing in the Simple trial. If the investigators will find an increased rate of findings (significantly higher than in the Simple trial ) it may set the stage for a randomized controlled trial of replacements , along the line of the Simple trial , or to a recommendation to continue VF testing in all ICD replacements.

DETAILED DESCRIPTION:
Background: The need for intraoperative defibrillation testing (DT) during implant and/ or replacement of implantable cardioverter-defibrillators (ICDs) is still in debate. The primary assumption of intra-operative DT is that successful defibrillation at the time of implant will predict successful treatment of clinical ventricular arrhythmias. However, the utility of this long standing practice in an era of modern very efficient ICD systems has recently been questioned. DT has not been proven to improve clinical outcomes, the relevance of test shocks to clinical shocks was questioned, and the probabilistic nature of successful shocks emphasized. Furthermore, testing may increase the risk, complexity and cost of ICD implants. This issue was addressed by the recent Shockless IMPLant Evaluation (SIMPLE) study. The trial demonstrated that routine defibrillation testing at the time of ICD implant was safe, but did not improve shock efficacy or reduce mortality compared to the no-testing strategy. It is therefore expected that the results of the SIMPLE trial will lead to a significant reduction or abandonment of the practice of VF testing at the time of initial ICD implant.

Nevertheless induction of VF for testing purposes (VFT) may still have an important role in selective populations that are at risk for defibrillation failure , who were not included in the SIMPLE study . One such population is of those who undergo device replacements. Whereas testing during replacement is seldom done , it is conceivable that this testing is going to have a much higher yield that during initial implantations . In fact, results from the Canadian ICD registry demonstrate a high rate of findings (up to 30%) when VF was induced during device replacements. However, it is conceivable that since most patients did not undergo testing, those were actually tested comprised a selected population with high likelihood of failure .

Testing at time of replacement has the potential to uncover lead problems specifically but not only in high voltage leads. Lovelock et al. have found that ICD generator replacement dramatically increased the risk of subsequent Fidelis lead failure and that the majority of these failures occurred within a matter of months after the procedure. Failure rates after generator replacement of other recalled or non- recalled leads are not known. It is possible that manipulation of the proximal portion of the lead during replacement or maybe clinically silent lead defects that were present prior to the generator exchange and that surgical manipulation accelerated the deterioration. Moreover, high energy shocks have been described to expose insulation defects not previously discovered by low energy shocks and noninvasive measurements.

Safety of DFT has also been a concern. The primary complications related to DT include: systemic embolism from intra-cardiac thrombus, prolonged post-DT hypotension and electro-mechanical dissociation, myocardial infarction, heart failure, cerebral anoxia, need for intubation, prolonged anesthesia, chest compressions and complications from anesthesia. The only large study to date which specifically evaluated this concern is the SIMPLE study. The primary safety endpoint, comprised of complications within 30 days of the implant, was also similar between the two patient groups (5.4 per cent )in the no-DT group vs. 6.5 per cent in the routine DT group, p=0.25). Thus, despite questions regarding the need for routine defibrillation testing, it is at least generally safe and may still be suitable for certain patients at the physician's discretion.

The SIMPLE study was a large one, and lasted quite a few years due to its design as a randomized controlled trial and the follow up needed to reach an endpoint. The investigators aim to conduct an observational pilot study looking at frequency of positive findings during VF testing . The comparator will be the rate of findings during testing in the Simple trial. If the investigators will find an increased rate of findings (significantly higher than in the Simple trial ) it may set the stage for a randomized controlled trial of replacements , along the line of the Simple trial , or to a recommendation to continue VF testing in all ICD replacements.

Study Objective:

The investigators plan to evaluate the rates of the following outcomes in subjects undergoing device replacement:

1. Failed DT
2. System malfunctions requiring intervention
3. Complications associated with DT during pocket generator change Secondary goals will include assessment of device longevity, specific ICD lead model performance , defibrillation efficacy, complications, association between replacement surgical techniques (i.e capsulectomy, electrosurgery settings and etc.) , data on lead management if failure was identified (adding a new lead, extraction and etc.) and rate of infection (i.e. association with type of antibiotics, IV vs PO, use of same pouch and etc.) The primary endpoint of this sub-study is a composite of procedure related complications including: 30-day procedure related infection, major bleeding ( (i.e prolonging hospital stay, reguiring intervention or PC units) new electrode dysfunction.

Study design:

This will be a prospective observational multi-center study of DF testing in all patients undergoing device replacement in the participating centers. All centers will follow the same DF testing protocol whereas management of positive findings will be at the discretion of the treating physicians, as will be the programming of devices following testing.

Primary Endpoint:

Demonstrate that the event rate of the primary outcome (defined as failure of DT at a single shock at 10 J below maximal capacity of the device

Secondary Endpoints:

The investigators plan to assess the following outcomes and determine independent predictors for their occurrence:

1. Rate of system malfunction requiring intervention
2. Complications associated with DT during pocket generator change.
3. Device longevity and specific ICD lead model performance
4. Lead management decisions in cases where lead failure is identified (adding a new lead, extraction and etc.)
5. Procedure related infections and opted management (i.e. association with type of antibiotics, IV vs. PO, use of same pouch and etc.)
6. Association between surgical replacement techniques (i.e capsulectomy, electrosurgery settings and etc.) and pre-specified complication rate

Patients will undergo generator replacement according to local procedure standards of practice. A minimum standard for VF evaluation will be a single shock at 10 J below maximal capacity of the device. If unsuccessful investigators are encouraged to use any appropriate method or testing to attain successful defibrillation. More extensive testing is permitted, if investigators deem it necessary. Investigators are free to use any method of anesthesia and patient monitoring that they feel is appropriate. All details of the operative procedure including if total or partial capsulectomy was done, DT conducted, intra-operative complications and device details will be captured at the time of implantation. The investigators will also collect data on longevity of device (time from implantation to replacement), use of antibiotics (IV and/or local, capsulectomy and use of plasma knife). Operators are encouraged to a high-voltage impedance test within the normal range of the device, to confirm the integrity of the high-voltage circuit in all patients. HV lead impedance will be documented. In cases of SJM Riata leads fluoroscopy of the lead will be done in LAO 30 and RAO 20 and documented.

VF testing : Patients will undergo induction of ventricular fibrillation (preferably Shock on T but will be left to operator discretion)during the implant procedure. For this study, a one shock at 10J below maximal device capacity will be programmed. If successful defibrillation is not achieved , it is recommended that all reasonable efforts should be made to achieve these criteria (i.e. addition of new lead/removal of coils or arrays, polarity reversal at operator discretion) followed by repeat intra-operative testing. Testing shall be stopped when the investigator deems that the likelihood of improving DFT by continued testing is outweighed by the risks. A reason for stopping shall be documented. Test shock will be done with new pocket generator and not old one.

Follow up: 6-monthly Follow-up visits: will include documentation of any peri-operative complications. Patients will be also followed for clinical endpoints (occurrence of appropriate shock, inappropriate shocks, lead failure, need for re- intervention and infection). Study visits will coincide as much as possible with routine clinical visits, allowing a flexibility of ± 1 month.

Patients will be followed at 6 monthly intervals until the last patient randomized has received 6 months of follow up.

Contact information (family physician, next of kin) will be obtained at baseline, and these individuals may be contacted during follow-up to ensure completeness of follow-up.

Sample Size Calculation: This is an observational study but in order to prove that replacements carry a higher risk of significant findings compared to primary implantations (as in the SIMPLE trial), the investigators will need 140 patients in order to detect an absolute difference of 7% in the rate of the primary endpoint (failure to terminated induced arrhythmia due to lead failure) with a power of 90% and 2-tailed alpha of 0.05 . This calculation is based on the estimation of 10% primary endpoint event rate in this study population that will be reported with a precision of ± 5%. Sample size calculation accounted for 10% overall attrition rate.

Budget was calculated by assumption of 500$ per patient fee for the participating centers plus study coordination and management costs.

The study will be managed by the Israeli Association for Cardiovascular Trials (IACT).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an ICD or CRT-D undergoing pocket generator replacement.

Exclusion Criteria:

1. If there is an absolute contraindication to DFT testing

   * NYHA class IV
   * AF > 24 hours unless on oral anticoagulation or negative TEE
   * Recent anoxic brain injury
2. Obvious lead malfunction (i.e. short V-V intervals, inappropriate shock for noise, clear fracture on CXR and etc.)
3. Unwilling to provide written informed consent
4. Unavailable for Follow-up
5. Pregnancy (or women of child-bearing potential not taking or willing to take an effective method of contraception).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an ICD or CRT-D undergoing pocket generator replacement.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-03 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Failure of DT at a single shock at 10 J below maximal capacity of the device | During replacement

SECONDARY OUTCOMES:
Rate of system malfunction requiring intervention | During procedure
Number of patients in which DT testing produced arrhythmia or ahock during procedure change | 6 month
Rate of lead failure or battery failure | 6 month
Lead management decisions in cases where lead failure is identified (adding a new lead, extraction and etc.) | During procedure
Number of patients with subsequent device infection and opted management (i.e. association with type of antibiotics, IV vs. PO, use of same pouch and etc.) | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Arrythmia Service Center, Ramat Gan, Israel